CLINICAL TRIAL: NCT04427215
Title: Effects of Complementary and Alternative Medicine on Mental Health in Breast Cancer Patients and Their Family Caregivers
Brief Title: Complementary and Alternative Medicine on Mental Health in Breast Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klaipėda University (Other)
Collaborators: Ministry of Health of The Republic of Lithuania (Unknown)
Responsible Party: Principal Investigator, Cesar Agostinis-Sobrinho, Principal Investigator, Klaipėda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: S-169
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Complementary Therapies

STUDY DESIGN:
Intervention Model Description: 5 intervention groups (music therapy, art therapy, dance-movement therapy, physical activity, bibliotherapy) and 1 control group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants will be randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A - Music Therapy (Experimental): Two section a week of music therapy
  Interventions: Other: Complementary and alternative medicines
- B - Art Therapy (Experimental): Two section a week of Art therapy
  Interventions: Other: Complementary and alternative medicines
- C - Dance-Movement Therapy (Experimental): Two section a week of Dance-Movement Therapy
  Interventions: Other: Complementary and alternative medicines
- D - Bibliotherapy (Experimental): Two section a week of Bibliotherapy
  Interventions: Other: Complementary and alternative medicines
- E - Physical Activity (Experimental): Two section a week of systematized physical activity
  Interventions: Other: Complementary and alternative medicines

INTERVENTIONS:
Other: Complementary and alternative medicines — Five types of Complementary and alternative medicines (Music Therapy, Art Therapy, Dance-Movement Therapy, Bibliotherapy, Physical Activity) will be applied twice a week.

SUMMARY:
During cancer treatment, several patient experience substantial psychological distress, mainly depression and anxiety, which can persist over years after completion of treatment.

Complementary and alternative medicine (CAM) has been in use among cancer patients for a long time and several types of CAM that are practiced in various parts of the world.

However, the effectiveness of different CAM therapies on mental health is still limited.

Therefore, the investigators want to assess the effectiveness of complementary and alternative medicine (CAM) (Dance/movement therapy, Art Therapy, Music Therapy, Bibliotherapy and Physical Activity) on mental health of cancer patients as well as their caregiver

DETAILED DESCRIPTION:
During cancer treatment, several patient experience substantial psychological distress, mainly depression and anxiety, which can persist over years after completion of treatment. These psychological impairments can aggravate symptom burden and can seriously affect health-related quality of life. Likewise, the diagnosis of cancer has not only a significant impact on the affected patients, but also on their families, and may cause emotional responses of shock, doubt, anxiety, and depression.

Complementary and alternative medicine (CAM) has been in use among cancer patients for a long time and several types of CAM that are practiced in various parts of the world. In the general among Lithuanian adult population, the use of CAM begins to seem common and the country claim for guidelines researches and to test the effectiveness of this practice to support the use of some CAM therapies on mental health of patients as well as their families.

In the St. Francis Oncology Center in Klaipeda some CAM have been applied aimed to increase the recovery and quality of life in the patients and their families. The effectiveness of different CAM therapies (Dance/movement therapy, Art Therapy, Music Therapy, Bibliotherapy and Physical Activity ) on mental health and recovery of cancer patients as well as on caregiving experiences and mental health of partners of cancer patients, it will be of great value to improve and provide a more effective service and the quality of caring in this patient as well as the continuing work of the Francis Oncology Center in Klaipeda and partners, with more higher scientific excellence and quality .

Objectives

· To assess the effectiveness of complementary and alternative medicine (CAM) (Dance/movement therapy, Art Therapy, Music Therapy, Bibliotherapy and Physical Activity) on mental health of cancer patients as well as their caregiver.

ELIGIBILITY:
Inclusion Criteria:

- All adult woman with breast cancer diagnoses and their primary family caregiver

Exclusion Criteria:

* Insufficient physical capacity
* Severe mental disorder
* Inability ti give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Mental Health | Mental health (score)changes over 4 weeks intervention
  Questionnaire to assess mental health
Quality of Life | Quality of life changes (score) over 4 weeks intervention
  Questionnaire to assess quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Cesar Agostinis-Sobrinho, Klaipėda, Lithuania

IPD SHARING:
Plan to Share IPD: No